CLINICAL TRIAL: NCT06260982
Title: Cognitive Disorders and Metabolism in 18-FDG- PET in Hereditary Spastic Paraplegia Type 4 (SPG4)
Brief Title: Cognitive Disorders in Hereditary Spastic Paraplegia Type 4
Acronym: SPG-TEP
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, RENAUD Mathilde, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2021PI148
Record Dates: First submitted 2023-06-26; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Spastic Paraplegia
Keywords: Hereditary Spastic Paraplegia type 4; 18-FDG-PET; cognitive disorders
MeSH Terms: conditions — Paraplegia; Cognitive Dysfunction | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: 18-FDG-PET — 18-FDG-PET and neuropsychological tests (language, memory, visuo-spatial tests, etc.).
  Other Names: neuropsychological testing

SUMMARY:
Hereditary spastic paraplegia type 4 is the most frequent mutation of hereditary spastic paraplegias. It is commonly described as pure, with progressive weakness of the lower limbs, pyramidal syndrome and vesico-sphincter disorders. However, cognitive disorders have been reported for over 20 years, but remain poorly characterized.

DETAILED DESCRIPTION:
Our primary objective is to describe a pattern of cognitive impairment in Hereditary Spastic Paraplegia type 4 using 18-FDG-PET metabolic imaging.

As secondary objectives, we wish to study the presence of correlations between neuropsychological tests, clinical examination, 18-FDG-PET data and general and genetic data of the pathology. We also wish to investigate correlations between genotype and phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age, living in the Grand Est region (France)
* Patient with a pathogenic or probably pathogenic variant (class 4 or 5) in the SPAST gene.

Exclusion Criteria:

* dementia comorbidities or cognitive disorders unrelated to the pathology that may affect neuropsychological tests.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed in the Grand Est region for type 4 spastic paraplegia with identification of a pathogenic or probably pathogenic variant in the SPAST gene.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01-02 (Estimated)

PRIMARY OUTCOMES:
cognitive testing | baseline
  we use detailed neuropsychological tests (MoCA)

SECONDARY OUTCOMES:
Correlations between neuropsychological tests, clinical examination, PET and general data. | baseline
Genotype/Phenotype correlations | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Renaud, Principal Investigator — Central Hospital Nancy
Locations (1):
- Centre hospitalier régional universitaire, Nancy, France